CLINICAL TRIAL: NCT00174356
Title: A Phase 1 Evaluation Of Oral CI-1033 In Combination With Paclitaxel And Carboplatin As First-Line Chemotherapy In Patients With Advanced Non-Small Cell Lung Cancer
Brief Title: PH 1 Evaluation Of Oral CI-1033 In Combination With Paclitaxel/ Carboplatin As 1st Line Chemotherapy In NSCLC Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A4161001
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2006-11-08 (Estimated); Status verified 2006-01

CONDITIONS: Carcinoma, Non-Small Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Canertinib; Paclitaxel; Carboplatin

INTERVENTIONS:
Drug: CI 1033
Drug: PACLITAXEL
Drug: CARBOPLATIN

SUMMARY:
The main purpose of this study is to evaluate the overall safety and maximum dose of CI 1033 in combination with paclitaxel and carboplatin in patients with NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* At least one target lesion that is unidimensionally measurable as defined by Response Evaluation Criteria in Solid Tumors (RECIST ; Appendix B.2 ) and has not been previously irradiated; a tumor that expresses at least one member of the erbB family of receptors (as determined by immunohistochemical evaluation by a Sponsor-designated core laboratory)

Exclusion Criteria:

* Prior chemotherapy, biologic therapy, immunotherapy, treatment with Herceptin, or treatment with investigational agents (including CI 1033); hormonal therapy within 28 days prior to baseline disease assessment (to exclude the possibility of a hormone-withdrawal response); prior definitive radiation therapy to the primary cancer site; not yet recovered from the acute effects of surgery or palliative radiotherapy; brain metastases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39
Dates: Start 2002-12; Study Completion 2005-10

PRIMARY OUTCOMES:
The primary objective is to evaluate the overall safety profile, including dose-limiting toxicities and the maximum tolerated dose, of CI 1033 in combination with paclitaxel (225 mg/m2) and carboplatin (area under the concentration time curve [AUC] of 6

SECONDARY OUTCOMES:
To determine the recommended Phase 2 dose of CI 1033 in combination with paclitaxel and carboplatin for patients with advanced NSCLC; to further define the safety profile of the recommended Phase 2 dose combination in an expanded cohort (22 patients)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (5):
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Park Ridge, Illinois
  - Pfizer Investigational Site, Skokie, Illinois
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Houston, Texas
- Pfizer Investigational Site, Hamilton, Ontario, Canada